CLINICAL TRIAL: NCT00724269
Title: Comparison of OPTI-FREE RepleniSH and ReNu Multi-Plus Lens Care Regimens on Corneal Epithelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: SMA-08-04 / BP-08-01
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2011-11

CONDITIONS: Contact Lens Wear
Keywords: Contact lens wear; multi-purpose solution; corneal staining

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opti Free RepliniSH (Active Comparator): Opti Free RepliniSH
  Interventions: Device: OPTI-FREE RepleniSH
- ReNu Multi-Plus (Active Comparator): ReNu Multi-Plus
  Interventions: Device: ReNu MultiPlus MPS

INTERVENTIONS:
Device: OPTI-FREE RepleniSH — Multi-Purpose Solution for soft contact lenses
  Arms: Opti Free RepliniSH
Device: ReNu MultiPlus MPS — Multi-Purpose Solution for soft contact lenses
  Arms: ReNu Multi-Plus

SUMMARY:
The purpose of this study is to evaluate the corneal epithelium after soft contact lens wear and use of two marketed multi-purpose solutions.

ELIGIBILITY:
Inclusion Criteria:

* Successful contact lens wear on a daily wear basis
* Wear contact lenses at least 8 hours/day
* Vision correctable to at least 20/30
* Normal Eyes
* Other protocol-defined inclusion criteria may apply

Exclusion:

* Topical ocular medication use
* Other protocol-defined inclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Confocal microscopy analysis of Corneal Epithelium | 2 weeks

SECONDARY OUTCOMES:
Patient comfort | 2 weeks
Corneal Staining | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Study Locations, Fort Worth, Texas, United States